CLINICAL TRIAL: NCT06671483
Title: A Multi-Center, Randomized, Double-Blind, Placebo- and Active-Controlled Phase 3 Study to Evaluate the Efficacy and Safety of Zasocitinib (TAK-279) in Subjects With Active Psoriatic Arthritis Who Are Naïve to Biologic Disease-Modifying Antirheumatic Drugs (LATITUDE-PsA-3001)
Brief Title: A Study of Zasocitinib in Adults With Psoriatic Arthritis Who Have Not Taken Biologic Medicines
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-279-PsA-3001; 2024-513111-27-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Psoriatic Arthritis
Keywords: Drug Therapy; Latitude Research Program; Latitude PsA; Latitude PsA-3001
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Zasocitinib Dose A (Experimental): Participants will receive zasocitinib Dose A, tablets, orally, once daily (QD) for up to Week 52.
  Interventions: Drug: Zasocitinib
- Zasocitinib Dose B (Experimental): Participants will receive zasocitinib Dose B, tablets, orally, QD for up to Week 52.
  Interventions: Drug: Zasocitinib
- Active Comparator Dose C (Active Comparator): Participants will receive active comparator Dose C, capsules, orally, twice daily (BID) for up to Week 52.
  Interventions: Drug: Active Comparator
- Placebo + Zasoctinib (Experimental): Participants will receive placebo, orally, QD for up to Week 16, followed by zasoctinib Dose A or Dose B, orally, QD, from Week 16 up to Week 52.
  Interventions: Drug: Zasocitinib; Drug: Placebo

INTERVENTIONS:
Drug: Zasocitinib — Zasocitinib over-encapsulated tablets.
  Other Names: TAK- 279; NDI-034858
  Arms: Placebo + Zasoctinib; Zasocitinib Dose A; Zasocitinib Dose B
Drug: Active Comparator — Active comparator capsule.
  Arms: Active Comparator Dose C
Drug: Placebo — Zasocitinib or active comparator matching placebo.
  Arms: Placebo + Zasoctinib

SUMMARY:
Psoriatic arthritis (PsA) is a chronic inflammatory disease that affects the joints and skin in people who have psoriasis (PsO).

The main aim of the study is to know how well zasocitinib (TAK-279) works in participants with active PsA who have not previously been treated with biologic disease-modifying antirheumatic drugs.

The participants will be treated with either zasocitinib, active comparator, or placebo. Participants will be in the study for up to 60 weeks.

ELIGIBILITY:
Inclusion Criteria:

Age:

1. The participant is aged 18 years or older at the time of signing the informed consent form (ICF). In South Korea, the age requirement for adult participants is >=19 years of age.

   Disease Characteristics:
2. The participant has a diagnosis of PsA.
3. The participant must have signs and symptoms of PsA for at least 3 months prior to screening.
4. The participant meets the Classification Criteria for Psoriatic Arthritis (CASPAR criteria).
5. The participant has active arthritis as shown by a minimum of >=3 tender joints in TJC68 and >=3 swollen joints in SJC66 at the screening and baseline (Day 1) visits.
6. The participant has at least 1 active lesion of plaque PsO >=2 cm in diameter, or any nail or nail bed changes characteristic of PsO.

   Medications for PsA:
7. The participant has had at least one of the following:

   1. Inadequate response to a nonsteroidal anti-inflammatory drug (NSAID) (not applicable in the European Union [EU]/ European Economic Area [EEA]), OR
   2. Inadequate response to a conventional synthetic disease-modifying antirheumatic drug (csDMARD).

Exclusion Criteria:

PsA and PsO:

1. The participant has other disease(s) that might confound the evaluations of benefit of zasocitinib therapy, including but not limited to rheumatoid arthritis, axial spondyloarthritis, systemic lupus erythematosus, Lyme disease, gout, or fibromyalgia.
2. The participant has a concomitant comorbid skin condition that, in the opinion of the investigator, would interfere with the study assessments, such as evidence of non-plaque PsO (erythrodermic, pustular, predominately guttate PsO, inverse, or drug-induced PsO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1088 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-05-18 (Estimated); Study Completion 2028-01-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving American College of Rheumatology 20 (ACR20) Response at Week 16 for Zasocitinib Dose A and B Compared to Placebo | At Week 16
  ACR responses are the numerical measurement of improvement in multiple disease assessment criteria. It is a composite clinical outcome assessment (COA) measure that includes both clinician-reported outcome assessments (ClinROs) and patient-reported outcomes (PROs). An ACR20 response is defined as: greater than or equal to (>=) 20 percent (%) improvement from baseline in both swollen joint count 66 joints (SJC66) and tender joint count 68 joints (TJC68), and >=20% improvement from baseline in 3 of the following 5 assessments: Patient's global assessment (PtGA) of psoriatic arthritis (PsA) pain; PtGA of PsA; physician's global assessment of disease activity (PGA) of PsA; participant's assessment of physical function as measured by health assessment questionnaire-disability index (HAQ-DI); high-sensitivity C-reactive protein (hsCRP). Percentage of participants achieving ACR20 response at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Minimal Disease Activity (MDA) at Week 16 for Zasocitinib Dose A and B Compared to Placebo | At Week 16
  The MDA is defined as a composite outcome measure of 7 ClinROs and PROs used in PsA. Participants are classified as achieving MDA if they fulfil 5 of 7 outcome measures: TJC68 less than or equal to (<=) 1, SJC66 <=1, psoriasis area and severity index (PASI) score <=1 or body surface area (BSA) affected by psoriasis <=3%, PtGA of PsA Pain score <=15, PtGA of PsA score <=20, HAQ-DI <=0.5, and Leeds Enthesitis Index (LEI) <=1. Percentage of participants achieving MDA at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Percentage of Participants Achieving PASI-75 Response (in Participants With a Baseline >=3% BSA) at Week 16 for Zasocitinib Dose A and B Compared to Placebo | Baseline, at Week 16
  A PASI-75 response is defined as >=75% improvement in the PASI score from baseline. It is a ClinRO used to measure psoriasis severity, combining the percent of affected skin surface area with the severity of erythema, induration, and desquamation across four body regions: head, upper extremities, trunk, and lower extremities. Severity is scored on a 0-4 scale, with 0 indicating no involvement and 4 indicating very marked involvement. PASI scores range from 0 to 72, with <=3 representing mild disease, >=3 to 15 representing moderate disease, and >=15 indicating severe disease. Percentage of participants achieving PASI-75 response (in participants with a baseline >=3% body surface area [BSA]) for zasocitinib Dose A and B compared to placebo at Week 16 will be reported.
Percentage of Participants Achieving ACR50 Response at Week 16 for Zasocitinib Dose A and B Compared to Placebo | At Week 16
  ACR responses are the numerical measurement of improvement in multiple disease assessment criteria. It is a composite COA measure that includes both ClinROs and PROs. An ACR50 response is defined as: >= 50% improvement from baseline in both SJC66 and TJC68, and >=50% improvement from baseline in 3 of the following 5 assessments: PtGA of PsA pain; PtGA of PsA; PGA of PsA; participant's assessment of physical function as measured by HAQ-DI; hsCRP. Percentage of participants achieving ACR50 response at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Change From Baseline in the HAQ-DI Score at Week 16 for Zasocitinib Dose A and B Compared to Placebo | Baseline, at Week 16
  The HAQ-DI is defined as a 20-item PRO measure used to assess functional ability over the past week across 8 categories: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. For each of these categories, participant reports the amount of difficulty they have in performing 2 or 3 specific activities on a 4-point scale (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, 3 = unable to do) The use of assistive devices and personal assistance are also noted. The HAQ-DI score is calculated as the mean of the category scores (0 = no disability, 3 = completely disabled), with 0 being the most desirable outcome and 3 as the least desirable. Participants must have scores for at least 6 categories for the HAQ-DI to be computed. Change from baseline in the HAQ-DI score at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Percentage of Participants Achieving ACR70 Response at Week 16 for Zasocitinib Dose A and B Compared to Placebo | At Week 16
  ACR responses are the numerical measurement of improvement in multiple disease assessment criteria. It is a composite COA measure that includes both ClinROs and PROs. An ACR70 response is defined as: >=70% improvement from baseline in both SJC66 and TJC68, and >=70% improvement from baseline in 3 of the following 5 assessments: PtGA of PsA pain; PtGA of PsA; PGA of PsA; participant's assessment of physical function as measured by HAQ-DI; hsCRP. Percentage of participants achieving ACR70 response at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Change From Baseline in the Short Form-36 Health Survey Version 2.0 (SF-36 v2.0) Physical Component Summary (PCS) Score at Week 16 for Zasocitinib Dose A Compared to Placebo | Baseline, at Week 16
  The SF-36 v2.0 is defined as a self-administered, validated questionnaire designed to measure general health-related quality of life (QoL). This 36-item questionnaire measures 8 domains over the past 4 weeks, including physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health, physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. Summary score PCS, will be calculated ranging from 0 (worst) to 100 (best). Higher scores indicate better QoL. Change from baseline in the SF-36 v2.0 PCS score at Week 16 for zasocitinib Dose A compared to placebo will be reported.
Change From Baseline in the Functional Assessment of Chronic Illness Therapy (FACIT)- Fatigue Score at Week 16 for Zasocitinib Dose A Compared to Placebo | Baseline, at Week 16
  The FACIT-fatigue score is defined as a 13-item PRO measure that assesses the severity of self-reported fatigue and its impact on daily functioning over the past 7 days. It includes items measuring tiredness, weakness, listlessness, lack of energy, and the effects on activities such as sleep and social interactions. Each item is rated on a 5-point scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; 4 = very much). The total score ranges from 0 to 52, with higher scores indicating less fatigue. Change from baseline in the FACIT- fatigue score at Week 16 for zasocitinib Dose A compared to placebo will be reported.
Percentage of Participants Achieving ACR20 Response at Week 16 for Zasocitinib Dose A and B Compared to Active Comparator | At Week 16
  ACR responses are the numerical measurement of improvement in multiple disease assessment criteria. It is a composite COA measure that includes both ClinROs and PROs. An ACR20 response is defined as: >= 20% improvement from baseline in both SJC66 and TJC68, and >=20% improvement from baseline in 3 of the following 5 assessments: PtGA of PsA pain; PtGA of PsA; PGA of PsA; participant's assessment of physical function as measured by HAQ-DI; hsCRP. Percentage of participants achieving ACR20 response of at Week 16 for zasocitinib Dose A and B compared to active comparator will be reported.
Percentage of Participants Achieving PASI-75 Response (in Participants With a Baseline >=3% BSA) at Week 16 for Zasocitinib Dose A compared to Active Comparator | Baseline, at Week 16
  A PASI-75 response is defined as >=75% improvement in the PASI score from baseline. It is a ClinRO used to measure psoriasis severity, combining the percent of affected skin surface area with the severity of erythema, induration, and desquamation across four body regions: head, upper extremities, trunk, and lower extremities. Severity is scored on a 0-4 scale, with 0 indicating no involvement and 4 indicating very marked involvement. PASI scores range from 0 to 72, with <=3 representing mild disease, >=3 to 15 representing moderate disease, and >=15 indicating severe disease. Percentage of participants achieving PASI-75 response (in participants with a baseline >=3% BSA) for zasocitinib Dose A compared to active comparator at Week 16 will be reported.
Percentage of Participants Achieving LEI =0 (in Participants With a Baseline LEI >=1) at Week 16 for Zasocitinib Dose A and B Compared to Placebo | Baseline, at Week 16
  The LEI is defined as a 6-item ClinRO measure specifically developed for PsA. It assesses the presence or absence of pain/tenderness when 4 kilograms per centimeter square (kg/cm^2) of pressure is applied to 6 enthesial sites: the lateral epicondyles, medial femoral condyles, and Achilles tendon insertions on both sides of the body. Tenderness at each site is recorded on a dichotomous scale (0 = non-tender, 1 = tender). The total score is the sum of tender sites, ranging from 0 to 6, with a higher score indicating a greater enthesitis burden. Percentage of participants achieving LEI =0 (in participants with a baseline LEI >=1) at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Change From Baseline in Individual Components of ACR Response at Week 16 for Zasocitinib Dose A and B Compared to Placebo | Baseline, at Week 16
  ACR responses are the numerical measurement of improvement in multiple disease assessment criteria. It is a composite COA measure that includes both ClinROs and PROs. An ACR response is defined as: improvement from baseline in both SJC66 and TJC68, and improvement from baseline in 3 of the following 5 assessments: PtGA of PsA pain (0-100 visual analogue scale [VAS]); PtGA of PsA (0-100 VAS); PGA of PsA (0-100 VAS); participant's assessment of physical function as measured by HAQ-DI (0-3 scale); hsCRP. Change from baseline in individual components of ACR response at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Percentage of Participants Achieving Leeds Dactylitis Index (LDI) =0 (in Participants With a Baseline LDI >=1) at Week 16 for Zasocitinib Dose A and B Compared to Placebo | Baseline, at Week 16
  The LDI is defined as a ClinRO measure use to assess the presence of dactylitis. It involves measuring the circumference of all 20 digits using a dactylometer, with measurements taken around the proximal phalanx as close to the web space as possible. Moderate pressure is applied to assess tenderness or pain in the affected digits. Tenderness is scored on a binary scale (0 = non-tender, 1 = tender). Only digits with a circumference ratio exceeding 10% are considered to have dactylitis. A higher score indicates worse dactylitis. Percentage of participants achieving LDI =0 (in participants with a baseline LDI >=1) at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Percentage of Participants Achieving PASI-75 Response (in Participants With a Baseline >=3% BSA) at Week 4 and 8 for Zasocitinib Dose A and B Compared to Placebo | Baseline, at Week 4 and 8
  A PASI-75 response is defined as >=75% improvement in the PASI score from baseline. It is a ClinRO used to measure psoriasis severity, combining the percent of affected skin surface area with the severity of erythema, induration, and desquamation across four body regions: head, upper extremities, trunk, and lower extremities. Severity is scored on a 0-4 scale, with 0 indicating no involvement and 4 indicating very marked involvement. PASI scores range from 0 to 72, with <=3 representing mild disease, >=3 to 15 representing moderate disease, and >=15 indicating severe disease. Percentage of participants achieving PASI-75 response (in participants with a baseline >=3% BSA) at Week 8 for zasocitinib Dose A and B compared to placebo will be reported.
Percentage of Participants Achieving PASI-90 Response (in Participants With a Baseline >=3% BSA) at Week 16 for Zasocitinib Dose A and B Compared to Placebo | Baseline, at Week 16
  A PASI-90 response is defined as >=90% improvement in the PASI score from baseline. It is a ClinRO used to measure psoriasis severity, combining the percent of affected skin surface area with the severity of erythema, induration, and desquamation across four body regions: head, upper extremities, trunk, and lower extremities. Severity is scored on a 0-4 scale, with 0 indicating no involvement and 4 indicating very marked involvement. PASI scores range from 0 to 72, with <=3 representing mild disease, >=3 to 15 representing moderate disease, and >=15 indicating severe disease. Percentage of participants achieving PASI-90 response (in participants with a baseline >=3% BSA) at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Percentage of Participants Achieving PASI-100 Response (in Participants With a Baseline >=3% BSA) at Week 16 for Zasocitinib Dose A and B Compared to Placebo | Baseline, at Week 16
  A PASI-100 response is defined as >=100% improvement in the PASI score from baseline. It is a ClinRO used to measure psoriasis severity, combining the percent of affected skin surface area with the severity of erythema, induration, and desquamation across four body regions: head, upper extremities, trunk, and lower extremities. Severity is scored on a 0-4 scale, with 0 indicating no involvement and 4 indicating very marked involvement. PASI scores range from 0 to 72, with <=3 representing mild disease, >=3 to 15 representing moderate disease, and >=15 indicating severe disease. Percentage of participants achieving PASI-100 response (in participants with a baseline >=3% BSA) at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Percentage of Participants Achieving ACR50 and PASI-100 Response (in Participants With a Baseline >=3% BSA) Simultaneously at Week 16 for Zasocitinib Dose A and B Compared to Placebo | Baseline, at Week 16
  ACR responses measure improvement in multiple criteria, a composite COA with ClinROs and PROs. An ACR50 response is >=50% improvement in SJC66 and TJC68, and 3 of 5 assessments: PtGA of PsA pain; PtGA of PsA; PGA of PsA, HAQ-DI, hsCRP. A PASI-100 response is >=100% improvement in the PASI score from baseline. It's a ClinRO measuring psoriasis severity, combining the percent of affected skin surface area with the severity of erythema, induration, and desquamation across four body regions: head, upper extremities, trunk, and lower extremities. Severity is scored from 0 (no involvement) to 4 (very marked involvement). PASI scores range from 0 to 72, with <=3 as mild, >=3 to 15 as moderate, and >=15 as severe disease. Percentage of participants achieving ACR50 and PASI-100 response (in participants with a baseline >=3% BSA) simultaneously at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Percentage of Participants Achieving sPGA Response of Clear (0) or Almost Clear (1) With >=2-Point Decrease From Baseline (in Participants With a Baseline sPGA >=2) at Week 16 for Zasocitinib Dose A and B Compared to Placebo | Baseline, at Week 16
  Static physician's global assessment (sPGA) is defined as a 5-point ClinRO measure used to assess the current state of psoriasis based on severity of erythema, induration, and scaling. The total sPGA score ranges from 0 to 4, where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe, with higher scores indicating greater disease severity. Each lesion characteristic (erythema, induration, and scaling) is graded separately on a 5-point scale: erythema (0 = no evidence to 4 = bright red coloration), induration (0 = no evidence to 4 = severe plaque elevation), and scaling (0 = no evidence to 4 = thick scaling). Lesion scores for erythema, induration, and scaling are averaged and rounded to nearest whole number to compute total score. Percentage of participants achieving sPGA response of clear (0) or almost clear (1) with >=2-point decrease from baseline (in participants with a baseline sPGA >=2) at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Percentage of Responders Achieving Minimal Clinically Important Differences (Reduction of >=0.35 From Baseline) in HAQ-DI Score From Baseline at Week 16 for Zasocitinib Dose A and B Compared to Placebo | Baseline, at Week 16
  The HAQ-DI is defined as a 20-item PRO measure used to assess functional ability over the past week across 8 categories: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Each category includes 2-3 activities rated on a 4-point scale (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, 3 = unable to do). Assistive devices and personal assistance are also noted. The HAQ-DI score is calculated as the mean of the category scores (0 = no disability, 3 = completely disabled), with scores of 0-1 indicating mild-to-moderate disability, 1-2 moderate-to-severe, and 2-3 severe-to-very severe disability. Participants must have scores for at least 6 categories for the HAQ-DI to be computed. Percentage of responders achieving minimal clinically important differences (reduction of >=0.35 from baseline) in HAQ-DI score from baseline at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Change From Baseline in the SF-36 v2.0 Mental Component Summary (MCS) Score at Week 16 for Zasocitinib Dose A and B Compared to Placebo | Baseline, at Week 16
  The SF-36 v2.0 is defined as a self-administered, validated questionnaire designed to measure general health-related quality of life (QoL). This 36-item questionnaire measures 8 domains over the past 4 weeks, including physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health, physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. Summary score MCS, will be calculated ranging from 0 (worst) to 100 (best). Higher scores indicate better QoL. Change from baseline in the SF-36 v2.0 MCS score at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Change From Baseline in Psoriatic Arthritis Impact of Disease-12 Items (PsAID-12) Total Score at Week 16 for Zasocitinib Dose A and B Compared to Placebo | Baseline, at Week 16
  The PsAID-12 is defined as a 12-item PRO measure that assesses symptoms such as pain, fatigue, and skin problems and the impact of PsA on the participant's life over the past week. It covers areas including work and/or leisure activities, physical activities, sleep, anxiety, embarrassment or shame, social participation, and depression. The response options are rated on a numerical rating scale (NRS) from 0 (none/no difficulty) to 10 (extreme difficulty), with higher scores indicating a greater impact of the disease. Change from baseline in PsAID-12 total score at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Change From Baseline in Disease Activity Index for Psoriatic Arthritis (DAPSA) Score at Week 16 for Zasocitinib Dose A and B Compared to Placebo | Baseline, at Week 16
  The DAPSA is defined as a composite measure of peripheral joint disease activity that includes ClinROs, PROs, and a laboratory test. DAPSA is calculated as the sum of the following components: tender joint count (0-68), swollen joint count (0-66), hsCRP level (milligrams per deciliter [mg/dL]), PtGA of PsA pain (0-100 VAS), and PtGA of PsA (0-100 VAS). DAPSA cutoffs for disease activity are: remission (<=4), low disease activity (>4 to <=14), moderate disease activity (>14 to <=28), and high disease activity (>28). Change from baseline in DAPSA score at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Change From Baseline in Disease Activity Score-28 (DAS28) (C-Reactive Protein) Score at Week 16 for Zasocitinib Dose A and B Compared to Placebo | Baseline, at Week 16
  The DAS28 with high-sensitivity C-reactive protein is defined as a derived index combining the tender joint count (28 joints), swollen joint count (28 joints), hsCRP, and PtGA of PsA. The 28-joint count includes the shoulder, elbow, wrist, metacarpophalangeal (MCP) 1-5, proximal interphalangeal (PIP) 1-5 of both upper extremities, and the knee joints of both lower extremities. The DAS28 score ranges from 0 to 10, with higher scores indicating greater disease activity. Change from baseline in DAS28 C-reactive protein score at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Change From Baseline in Physician's Global Assessment of Fingernail Psoriasis (PGA-F) Score in Participants With Psoriatic Nail Involvement (PGA-F Greater than [>] 0) From Baseline at Week 16 for Zasocitinib Dose A and B Compared to Placebo | Baseline, at Week 16
  The PGA-F is defined as a ClinRO measure assessing the severity of fingernail PsO. It evaluates nail bed signs (onycholysis, hyperkeratosis, erythema, splinter hemorrhages) and nail matrix signs (pitting, ridging, discoloration). Clinicians rate the severity using categories: clear (0), minimal (1), mild (2), moderate (3), and severe (4). The total score is based on the area with the most involvement (nail bed or matrix), ranging from 0 (clear) to 4 (very severe), with higher scores indicating more severe fingernail PsO. Change from baseline in PGA-F score in participants with PGA-F >0 from baseline at Week 16 for zasocitinib Dose A and B compared to placebo will be reported.
Percentage of Participants Achieving a Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesis Index = 0 through Week 16 for Zasocitinib Dose A and B Compared to Placebo | Baseline up to Week 16
  The SPARCC Enthesis Index is a ClinRO measure that assesses the presence or absence of pain/tenderness when 4 kg/cm^2 of pressure is applied to 18 enthesial sites across the following 9 bilateral sites: Achilles tendons, plantar fascia insertion at the calcaneus, greater tuberosity of the humerus, medial epicondyles, lateral epicondyles, greater trochanter, quadriceps insertion, inferior patella, and tibial tuberosity. Tenderness at each site is recorded as either present (1) or absent (0). Total score is the sum of score from each site, ranging from 0 to 16, with higher scores indicating greater enthesis burden. Percentage of participants achieving SPARCC Enthesis Index = 0 through Week 16 for zasocitinib Dose A and B compared to placebo will be reported
Percentage of Participants Achieving ACR20 Response at Week 8 for Zasocitinib Dose A and B Compared to Placebo | At Week 8
  ACR responses are the numerical measurement of improvement in multiple disease assessment criteria. It is a composite COA measure that includes both ClinROs and PROs. An ACR20 response is defined as: >= 20% improvement from baseline in both SJC66 and TJC68, and >=20% improvement from baseline in 3 of the following 5 assessments: PtGA of PsA pain; PtGA of PsA; PGA of PsA; participant's assessment of physical function as measured by HAQ-DI; hsCRP. Percentage of participants achieving ACR20 response at Week 8 for zasocitinib Dose A and B compared to placebo will be reported.
Change From Baseline in the SF-36 v2.0 PCS Score at Week 16 for Zasocitinib Dose B Compared to Placebo | Baseline, at Week 16
  The SF-36 v2.0 is defined as a self-administered, validated questionnaire designed to measure general health-related quality of life (QoL). This 36-item questionnaire measures 8 domains over the past 4 weeks, including physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health, physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. Summary score PCS, will be calculated ranging from 0 (worst) to 100 (best). Higher scores indicate better QoL. Change from baseline in the SF-36 v2.0 PCS score at Week 16 for zasocitinib Dose B compared to placebo will be reported.
Change From Baseline in the FACIT- Fatigue Score at Week 16 for Zasocitinib Dose B Compared to Placebo | Baseline, at Week 16
  The FACIT-fatigue score is defined as a 13-item PRO measure that assesses the severity of self-reported fatigue and its impact on daily functioning over the past 7 days. It includes items measuring tiredness, weakness, listlessness, lack of energy, and the effects on activities such as sleep and social interactions. Each item is rated on a 5-point scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; 4 = very much). The total score ranges from 0 to 52, with higher scores indicating less fatigue. Change from baseline in the FACIT- fatigue score at Week 16 for zasocitinib Dose B compared to placebo will be reported.
Percentage of Participants Achieving ACR50 Response at Week 16 for Zasocitinib Dose A and B Compared to Active Comparator | At Week 16
  ACR responses are the numerical measurement of improvement in multiple disease assessment criteria. It is a composite COA measure that includes both ClinROs and PROs. An ACR50 response is defined as: >= 50% improvement from baseline in both SJC66 and TJC68, and >=50% improvement from baseline in 3 of the following 5 assessments: PtGA of PsA pain; PtGA of PsA; PGA of PsA; participant's assessment of physical function as measured by HAQ-DI; hsCRP. Percentage of participants achieving ACR50 response at Week 16 for zasocitinib Dose A and B compared to active comparator will be reported.
Percentage of Participants Achieving ACR70 Response at Week 16 for Zasocitinib Dose A and B Compared to Active Comparator | At Week 16
  ACR responses are the numerical measurement of improvement in multiple disease assessment criteria. It is a composite COA measure that includes both ClinROs and PROs. An ACR70 response is defined as: >=70% improvement from baseline in both SJC66 and TJC68, and >=70% improvement from baseline in 3 of the following 5 assessments: PtGA of PsA pain; PtGA of PsA; PGA of PsA; participant's assessment of physical function as measured by HAQ-DI; hsCRP. Percentage of participants achieving ACR70 response at Week 16 for zasocitinib Dose A and B compared to active comparator will be reported.
Percentage of Participants Achieving PASI-90 Response (in Participants With a Baseline >=3% BSA) at Week 16 for Zasocitinib Dose A and B Compared to Active Comparator | Baseline, at Week 16
  A PASI-90 response is defined as >=90% improvement in the PASI score from baseline. It is a ClinRO used to measure psoriasis severity, combining the percent of affected skin surface area with the severity of erythema, induration, and desquamation across four body regions: head, upper extremities, trunk, and lower extremities. Severity is scored on a 0-4 scale, with 0 indicating no involvement and 4 indicating very marked involvement. PASI scores range from 0 to 72, with <=3 representing mild disease, >=3 to 15 representing moderate disease, and >=15 indicating severe disease. Percentage of participants achieving PASI-90 response (in participants with a baseline >=3% BSA) at Week 16 for zasocitinib Dose A and B compared to active comparator will be reported.
Percentage of Participants Achieving PASI-100 Response (in Participants With a Baseline >=3% BSA) at Week 16 for Zasocitinib Dose A and B Compared to Active Comparator | Baseline, at Week 16
  A PASI-100 response is defined as >=100% improvement in the PASI score from baseline. It is a ClinRO used to measure psoriasis severity, combining the percent of affected skin surface area with the severity of erythema, induration, and desquamation across four body regions: head, upper extremities, trunk, and lower extremities. Severity is scored on a 0-4 scale, with 0 indicating no involvement and 4 indicating very marked involvement. PASI scores range from 0 to 72, with <=3 representing mild disease, >=3 to 15 representing moderate disease, and >=15 indicating severe disease. Percentage of participants achieving PASI-100 response (in participants with a baseline >=3% BSA) at Week 16 for zasocitinib Dose A and B compared to active comparator will be reported.
Percentage of Participants Achieving ACR50 and PASI-100 Response (in Participants With a Baseline >=3% BSA) Simultaneously at Week 16 for Zasocitinib Dose A and B Compared to Active Comparator | Baseline, at Week 16
  ACR responses measure improvement in multiple criteria, a composite COA with ClinROs and PROs. An ACR50 response is >=50% improvement in SJC66 and TJC68, and 3 of 5 assessments: PtGA of PsA pain; PtGA of PsA; PGA of PsA, HAQ-DI, hsCRP. A PASI-100 response is >=100% improvement in the PASI score from baseline. It's a ClinRO measuring psoriasis severity, combining the percent of affected skin surface area with the severity of erythema, induration, and desquamation across four body regions: head, upper extremities, trunk, and lower extremities. Severity is scored from 0 (no involvement) to 4 (very marked involvement). PASI scores range from 0 to 72, with <=3 as mild, >=3 to 15 as moderate, and >=15 as severe disease. Percentage of participants achieving ACR50 and PASI-100 response (in participants with a baseline >=3% BSA) simultaneously at Week 16 for zasocitinib Dose A and B compared to active comparator will be reported.
Percentage of Participants Achieving Minimal Disease Activity (MDA) at Week 16 for Zasocitinib Dose A and B Compared to Active Comparator | At Week 16
  The MDA is defined as a composite outcome measure of 7 ClinROs and PROs used in PsA. Participants are classified as achieving MDA if they fulfil 5 of 7 outcome measures: TJC68 less than or equal to (<=) 1, SJC66 <=1, psoriasis area and severity index (PASI) score <=1 or body surface area (BSA) affected by psoriasis <=3%, PtGA of PsA Pain score <=15, PtGA of PsA score <=20, HAQ-DI <=0.5, and Leeds Enthesitis Index (LEI) <=1. Percentage of participants achieving MDA at Week 16 for zasocitinib Dose A and B compared to active comparator will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (195):
- United States (53):
  - AARR- Chandler AZ, Chandler, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC | Phoenix, AZ, Phoenix, Arizona
  - First OC Dermatology Research Inc., Fountain Valley, California
  - Purushotham & Akther Kotha MD, La Mesa, California
  - Triwest Research Associates LLC, La Mesa, California
  - VA Northern California Health Care System - NAVREF - PPDS, Mather, California
  - Biosolutions Research Center | La Mesa, CA, Poway, California
  - The Cohen Medical Centers, Thousand Oaks, California
  - Foothill Arthritis Clinic, Tujunga, California
  - Medvin Clinical Research, Whittier, California
  - Denver Arthritis Clinic | Denver, CO, Denver, Colorado
  - Arthritis & Rheumatic Disease Specialties (AARDS), Aventura, Florida
  - RASF- Clinical Research Center, Boca Raton, Florida
  - Clinical Research of West Florida | Clearwater, FL, Clearwater, Florida
  - GNP Research, LLC | Hollywood, FL, Cooper City, Florida
  - Driven Research LLC, Coral Gables, Florida
  - Tectum Medical Research, Davie, Florida
  - Sweet Hope Research Specialty, Inc, d/b/a Neoclinical Research, Hialeah, Florida
  - Bioresearch Partners, Miami, Florida
  - HMD Research LLC, Orlando, Florida
  - Millennium Research | Ormond Beach, FL, Ormond Beach, Florida
  - IRIS Research and Development | Plantation, FL, Plantation, Florida
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - West Broward Rheumatology Associates, Inc., Tamarac, Florida
  - Clinical Research of West Florida | Tampa, FL, Tampa, Florida
  - Marietta Rheumatology Associates, Marietta, Georgia
  - GSCP/CIS, Orland Park, Illinois
  - Greater Chicago Specialty Physicians LLC/CIS, Schaumburg, Illinois
  - Accurate Clinical Research, Inc. | Lake Charles, Lake Charles, Louisiana
  - Klein & Associates, M.D., P.A., Hagerstown, Maryland
  - Henry Ford Health System-Rheumatology Department, Detroit, Michigan
  - Michigan Rheumatology Group, P.C. - Grand Blanc Office, Grand Blanc, Michigan
  - Ash Research Clinic - Howell, Howell, Michigan
  - June DO, PC Private Practice - Dr. Justus Fiechtner, Lansing, Michigan
  - Clinical Research Institute of Michigan, Saint Clair Shores, Michigan
  - Saint Louis Rheumatology, St Louis, Missouri
  - Albuquerque Center for Rheumatology PC, Albuquerque, New Mexico
  - Santa Fe Rheumatology, Santa Fe, New Mexico
  - NYU Langone Health | Joseph S. and Diane H. Steinberg Ambulatory Care Center - Rheumatology Department, Brooklyn, New York
  - Accellacare of Hickory, Hickory, North Carolina
  - University Hospitals | UH Cleveland Medical Center - Department of Medicine - Rheumatology Division, Cleveland, Ohio
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - PA Regional Center for Arthritis and Osteoporosis Research, Wyomissing, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - Accurate Clinical Research, Baytown, Texas
  - Novel Research | Bellaire Location, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Introscience Research | Northwest Houston Arthritis Center - Houston, TX, Houston, Texas
  - West Texas Clinical Research, Lubbock, Texas
  - Southwest Rheumatology Research, LLC | Mesquite, TX, Mesquite, Texas
  - Clinical Investigations of Texas, Plano, Texas
  - Arthritis Northwest, PLLC | Spokane, WA, Spokane, Washington
  - Medical College of Wisconsin | Department of Medicine - Rheumatology Division, Milwaukee, Wisconsin
- Belgium (5):
  - Université Libre de Bruxelles, Anderlecht, Brussels Capital
  - University Hospital Ghent, Ghent, Flanders
  - ReumaClinic Genk, Genk, Limburg
  - St Pierre Brussels, Brussels
  - Centre Hospitalier Universitaire (CHU) de Liege - Domaine Universitaire du Sart Tilman, Liège
- Bulgaria (9):
  - Diagnostic Consultative Centre - Focus-5 - LZIP EOOD, Sofia, Sofia-Grad
  - Military Medical Academy Multiprofile Hospital for Not Yet Recruiting Treatment - Sofia, Sofia, Sofia-Grad
  - Centre of Rheumatology St. Irina, Sofia, Sofia-Grad
  - Medical Center Medconsult Pleven OOD, Pleven
  - AES Partner Site -Plovdiv, Plovdiv
  - Medical Center Artmed OOD | Plovdiv, Bulgaria, Plovdiv
  - Diagnostic- Consultative Center- 1- Ruse EOOD, Rousse
  - Dr Stoyanka Vladeva IPSMP VBR | Stara Zagora, Bulgaria, Stara Zagora
  - Medical Center Zara-Med EOOD, Stara Zagora
- Chile (5):
  - El Centro de Estudios Reumatologicos (CER), Providencia, Santiago Metropolitan
  - Clinica Dermacross S.A., Santiago, Santiago Metropolitan
  - Centro de Estudios Clinicos, Santiago
  - CTR Estudios, Santiago
  - Centro Internacional de Estudios Clínicos, Santiago
- Colombia (5):
  - Centro Integral de Reumatologia Circaribe S.A.S., Barranquilla, Atlántico
  - Centro de Investigacion en Reumatologia y Especialidades Medicas S.A.S, CIREEM S.A.S, Bogota D.C., Cundinamarca
  - Fundacion Santa Fe de Bogota, Bogotá D.C., Cundinamarca
  - Servimed S.A.S, Bucaramanga, Cundinamarca
  - Preventive Care S.A.S., Chía, Cundinamarca
- Croatia (5):
  - Medicinski Centar Kuna and Peric, Zagreb, City of Zagreb
  - Clinical Hospital Centre Osijek, Osijek
  - Clinical Hospital Center Rijeka, Rijeka
  - University Hospital Centre Split, Split
  - General Hospital Zadar, Zadar
- Czechia (9):
  - Revmatologie s.r.o. | Brno, Czech Republic, Brno, Czech Rep
  - L.K.N. Arthrocentrum, s.r.o. - Revmatologicka, Hlučín, Czech Rep
  - Clintrial s.r.o. | Prague, Czech Republic, Prague, Czech Rep
  - Praglandia | Prague, Czech Republic, Prague, Czech Rep
  - MEDICAL Plus s.r.o., Uherské Hradiště, Czech Rep
  - CCR Ostrava, Ostrava, Moravskoslezský kraj
  - Pv Medical Services, Zlín, NAP
  - Revmatologicky ustav | Clinical Evaluation Department, Prague, Prague
  - Pratia Pardubice a.s., Pardubice
- Estonia (5):
  - Innomedica OU | Tallinn, Estonia, Tallinn, Harju
  - Center for Clinical and Basic Research, Tallinn, Harju
  - Clinical Research Centre | Tartu, Estonia, Tartu, Tartu
  - North Estonia Medical Centre | Mustamae Building - Internal Medicine Clinic - Rheumatology Department, Tallinn
  - MediTrials OÜ, Tartu
- Germany (8):
  - Fachklinik Bad Bentheim, Bad Bentheim, Lower Saxony
  - Rheumzentrum Prof.Dr.med.Gunther Neeck, Bad Doberan, Mecklenburg-Vorpommern
  - Rheumazentrum Ratingen-Studienambulanz, Ratingen, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig AoeR, Leipzig, Saxony
  - Rheumatologische Schwerpunktpraxis | Berlin, Germany, Berlin
  - Städtisches Klinikum Dresden, Dresden
  - MVZ Rheumatologie und Autoimmunmedizin Hamburg GmbH - Hamburg, Hamburg
  - Medicover MVZ München Ost, München
- Hungary (6):
  - Porcika Klinika, Hódmezővásárhely, Csongrad-Csanad
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged, Csongrad-Csanad
  - CMed Rehabilitacios es Diagnosztikai Kozpont, Székesfehérvár, Fejér
  - Qualiclinic | Budapest, Hungary, Budapest
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktató Korhaz | Rheumatology Department - Arthritis Center, Székesfehérvár
  - Vital Medical Center Medical Center and Dental Center | Reumatologia - Veszprem, Hungary, Veszprém
- Israel (6):
  - Assuta Ashdod Medical Center, Ashdod, Southern District
  - Barzilai Medical Center | Rheumatology Department, Ashkelon
  - Rambam Health Care Campus, Haifa
  - Galilee Medical Center | Rheumatology Unit, Nahariya
  - The Chaim Sheba Medical Center - The Zabludowicz Center for Autoimmune Diseases, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (9):
  - Azienda Ospedaliero-Universitaria delle Marche; SOD Clinica Medica, Torrette, Ancona
  - Fondazione PTV Policlinico Tor Vergata, Rome, Lazio
  - Policlinico Agostino Gemelli, UOC Reumatology, Rome, Lazio
  - ASST Centro Specialistico Ortopedico Traumatologico Gaetano Pini-CTO, Milan, Lombardy
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele, Milan, Lombardy
  - IRCCS Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedale Università Padova, Padua, Veneto
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Latvia (2):
  - D. Saulites Kandevicas Private Practice in Cardiology and Rheumatology | Liepaja, Latvia, Liepāja
  - ORTO Clinic | Rheumatology Department, Riga
- Mexico (10):
  - Centro de Investigacion en Artritis y Osteoporosis S.C. (CIAO), Mexicali, Estado de Baja California
  - iBiomed Guadalajara, Zapopan, Guadalajara
  - Centro Integral en Reumatologia, S.A. de C.V., Guadalajara, Jalisco
  - Private Practice - Dr. Delfina Villanueva Quintero, Guadalajara, Jalisco
  - Consultorio de Reumatologia, Gustavo Adolfo Madero, Mexico City
  - HMG Hospital Coyoacan, Mexico City, Mexico City
  - CINTRE, Centro de Investigacion y Tratamiento Reumatologico S.C., Mexico City, Mexico City
  - Kohler and Milstein Research Yucatan, Mérida, Yucatán
  - Hospitales Star Medica, Mérida, Yucatán
  - Office of Cesar F. Pacheco-Tena, MD, Chihuahua City
- New Zealand (5):
  - CGM Research Trust, Christchurch Central, Christchurch
  - Aotearoa Clinical Trials, Auckland, North Island
  - North Shore Hospital, Auckland, North Island
  - Porter Rheumatology Ltd, Nelson, South Island
  - Waikato Hospital, Hamilton, Waikato Region
- Poland (28):
  - Pratia Poznań, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne Plejady, Krakow, Lesser Poland Voivodeship
  - Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship
  - Krakowskie Centrum Medyczne, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Katowice - PRATIA, Katowice, Lower Silesian Voivodeship
  - WroMedica Centrum Zdrowia | Rheumatology Clinic, Wroclaw, Lower Silesian Voivodeship
  - RCMed | Sochaczew, Poland, Sochaczew, Masovian Voivodeship
  - Rheuma Medicus | Warsaw, Poland, Warsaw, Masovian Voivodeship
  - MTZ Clinical Research Powered by PRATIA, Warsaw, Masovian Voivodeship
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. prof. dr hab. med. Eleonory Reicher, Centrum Wsparcia Badań Klinic, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Reuma Park, Warsaw, Masovian Voivodeship
  - ETG Warszawa Sp. z o.o., Warsaw, Masovian Voivodeship
  - Twoja Przychodnia Opolskie Centrum Medyczne, Opole, Opole Voivodeship
  - INTER CLINIC Piotr Adrian Klimiuk | Bialystok, Poland, Bialystok, Podlaskie Voivodeship
  - Nova Reuma Domyslawska i Rusilowicz- Spolka Partnerska Lekarza Reumatologa i Fizjoterapeuty, Bialystok, Podlaskie Voivodeship
  - Zdrowie Osteo Medic sc L i A Racewicz, A i J Supronik, Bialystok, Podlaskie Voivodeship
  - Bif-Med s.c. NZOZ, Bytom, Silesian Voivodeship
  - MICS Centrum Medyczne Torun, Torun, Silesian Voivodeship
  - UNICA CR sp. z.o. o., Dąbrówka, Warmian-Masurian Voivodeship
  - Ambulatorium Sp. z o.o., Elblag, Warmian-Masurian Voivodeship
  - Etyka Osrodek Badan Klinicznych | Olsztyn, Poland, Olsztyn, Warmian-Masurian Voivodeship
  - Twoja Przychodnia - Poznanskie Centrum Medyczne Sp. z o.o., Poznan, Wielkopolska
  - Reumedika | Poznan, Poland, Poznan, Wlkp
  - Prywatna Praktyka Lekarska Prof. dr hab. med. Pawel Hrycaj | Poznan, Poland, Poznan, Woj. Wielkopolskie
  - Santa Familia PTG Lodz | Lodz, Poland, Lodz
  - FutureMeds | Lodz Center - Lodz, Poland, Lodz
  - Twoja Przychodnia | Nowa Sol, Poland, Nowa Sól
  - FutureMeds Wroclaw, Wroclaw
- Portugal (7):
  - Centro Hospitalar e Universitário de Coimbra E.P.E - Hospitais da Universidade de Coimbra, Coimbra, Barcelona
  - Hospital Conde de Bertiandos Unidade Local de Saúde Do Alto Minho, Ponte de Lima, Barcelona
  - Centro Hospitalar de Vila Nova de Gaia / Espinho E.P.E, Vila Nova de Gaia, New Mexico
  - Hospital Garcia de Orta, Almada
  - Centro Hospitalar e Universitário de Coimbra E.P.E - Hospitais da Universidade de Coimbra, Coimbra
  - Instituto Portugues de Reumatologia, Lisbon
  - Centro Hospitalar Universitario de Lisboa Norte | Hospital Santa Maria - Rheumatology Department, Lisbon
- Puerto Rico (2):
  - Centro Reumatologico de Caguas | Caguas, PR, Caguas
  - GCM Medical Group, PSC | San Juan, PR, San Juan
- South Korea (5):
  - The Catholic University of Korea, Suwon, Gyeonggi-do
  - Ajou University Hospital | Clinical Trial Center, Suwon, Gyeonggido
  - Asan Medical Center, Seoul
  - SMG - SNU Boramae Medical Center, Seoul
  - Kyung Hee University Hospital, Seoul
- Spain (6):
  - Hospital Universitario de Badajoz, Mérida, Badajoz
  - Corporacio Sanitaria Parc Tauli - Hospital de Sabadell, Sabadell, Barcelona
  - Hospital Clinico Universitario de Santiago de Compostela | Building A - Rheumatology Department, Santiago de Compostela, Galicia
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (5):
  - National Cheng Kung University, Tainan, Tainan City
  - National Taiwan University Hospital, Zhong Zheng Qu, Taipei City
  - Far Eastern Memorial Hospital | Allergy, Immunology and Rheumatology Department, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - Chi Mei Medical Center, Tainan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/175345f32479452b